CLINICAL TRIAL: NCT06140823
Title: Prospective Validation of Liver Cancer Risk Computation (LIRIC) Models on Multicenter EHR Data
Brief Title: Prospective Validation of Liver Cancer Risk Computation (LIRIC) Models
Status: Active, not recruiting | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Massachusetts Institute of Technology (Other); TriNetX, LLC (Unknown)
Responsible Party: Principal Investigator, Limor Appelbaum, Principal Investigator, Beth Israel Deaconess Medical Center
Other Study IDs: Nov2023Trial
Record Dates: First submitted 2023-11-15; First posted 2023-11-20 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Predictive Cancer Model

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- prospective general population cohort: Males and females age >= 40 years, without a personal history of HCC or current HCC and at least two clinical visits to their HCO, within the last year, before the study start date.
  Interventions: Other: Liver Risk Computation Model (LIRIC)
- Prospective cirrhosis population cohort: Males and females age >= 40 years, with liver cirrhosis and without a personal history of HCC or current HCC, that have at least two clinical visits to their HCO, within the last year, before the study start date.
  Interventions: Other: Liver Risk Computation Model (LIRIC)_cirrhosis
- Prospective no_cirrhosis population cohort: Males and females age >= 40 years, without a personal history of HCC or current HCC and without a diagnosis of liver cirrhosis, that have at least two clinical visits to their HCO, within the last year, before the study start date.
  Interventions: Other: Liver Risk Computation Model (LIRIC)_no_cirrhosis

INTERVENTIONS:
Other: Liver Risk Computation Model (LIRIC) — A neural network model (LIRIC-NN) and a logistic regression model (LIRIC-LR) that use routinely collected EHR data to stratify individuals into HCC risk groups for the general population
  Groups: prospective general population cohort
Other: Liver Risk Computation Model (LIRIC)_cirrhosis — A neural network model (LIRIC-NN) and a logistic regression model (LIRIC-LR) that use routinely collected EHR data to stratify individuals into HCC risk groups for the population with liver cirrhosis
  Groups: Prospective cirrhosis population cohort
Other: Liver Risk Computation Model (LIRIC)_no_cirrhosis — neural network model (LIRIC-NN) and a logistic regression model (LIRIC-LR) that use routinely collected EHR data to stratify individuals into HCC risk groups for the population without liver cirrhosis
  Groups: Prospective no_cirrhosis population cohort

SUMMARY:
The goal of this prospective observational cohort study is to validate previously developed Hepatocellular Carcinoma (HCC) risk prediction algorithms, the Liver Risk Computation (LIRIC) models, which are based on electronic health records.

The main questions it aims to answer are:

* Will our retrospectively developed general population LIRIC models, developed on routine EHR data, perform similarly when prospectively validated, and reliably and accurately predict HCC in real-time?
* What is the average time from model deployment and risk prediction, to the date of HCC development and what is the stage of HCC at diagnosis?

The risk model will be deployed on data from individuals eligible for the study. Each individual will be assigned a risk score and tracked over time to assess the model's discriminatory performance and calibration.

DETAILED DESCRIPTION:
The investigators will conduct a prospective observational cohort study, separately deploying three separate LIRIC models (the general population, cirrhosis, and no_cirrhosis models) on retrospective de-identified EHR data of 44 HCOs in the USA, using the TriNetX federated network platform. LIRIC will generate a risk score for each individual. All risk-stratified individuals will be prospectively, electronically followed for up to 3-years to assess the primary end-point of HCC development. At the end of this period, model discrimination will be assessed, using the following metrics: AUROC, sensitivity, specificity, PPV/NPV. Risk scores generated by the model will be divided into quantiles. For each quantile, the investigators will evaluate the following: number of individuals in each quantile, number of HCC cases, PPV, NNS, SIR. Model calibration will be used for assessing the accuracy of estimates, based on the estimated to observed number of events. The model will dynamically re-evaluate all individual data every 6 months, re-classifying individuals (as needed).

ELIGIBILITY:
The investigators will utilize the following criteria for all 3 models:

Inclusion criteria:

* Male and females age ≥40 years from all US HCOs available on the platform
* at least at least 2 clinical encounters to the HCO, within the last year, before the study start date

Exclusion Criteria:

* Personal history of HCC or current HCC (ICD-9: 155.0; ICD-10: C22.0)
* Age below 40. The same dataset will be utilized for the non-cirrhosis validation, with exclusion of all cases with cirrhosis (ICD-9: 571.2, 571.5; ICD-10: K70, K70.3, K70.30, K70.31, K74, K74.0, K74.6, K74.60, K74.69). For the cirrhosis validation, the investigators will include only patients with the above cirrhosis codes.

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The cohort will be selected from 44 eligible HCOs comprised of community hospitals, outpatient clinics and academic medical centers from across the US.
Sampling Method: Non-Probability Sample
Enrollment: 6000000 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Area under the receiver operating characteristic curve (AUROC) of LIRIC for all groups stratified | 6 months from index date, at 1 year, 2 years and 3 years
  To assess the discriminatory performance of LIRIC for prospective identification of high-risk individuals for HCC development. ROCs and AUROC numbers will be calculated for the whole population and groups stratified by age, sex, race, and geographical location.
Calibration of LIRIC for all groups stratified | 6 months from index date, at 1 year, 2 years and 3 years
  To assess how well the risk prediction by LIRIC aligns with observed risk without recalibration. Calibration plots will be created for the whole population and groups stratified by age, sex, race, and geographical location.
Performance metrics for LIRIC model risk quantiles | 6 months from index date, at 1 year, 2 years and 3 years
  To evaluate the sensitivity, specificity, number of individuals/number of HCC cases, PPV, NNS in each predicted risk quantile for multiple risk thresholds

SECONDARY OUTCOMES:
Timing of incident HCC occurrence | 6 months from index date, at 1 year, 2 years and 3 years
  To evaluate how long in advance before HCC occurrence should be expected for LIRIC models to make high-risk predictions based on different thresholds for high-risk. Distribution plots of the date of HCC incidence for multiple risk thresholds will be created.
Tumor stage at HCC diagnosis | 6 months from index date, at 1 year, 2 years and 3 years
  TNM staging at HCC diagnosis

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States